CLINICAL TRIAL: NCT05272449
Title: Evaluation of a Disposable Sound Sensor for Recording Respiration During Sleep
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CIDELEC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-A02524-37
Record Dates: First submitted 2022-02-17; First posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Sleep Apnea (Disorder)
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation of a disposable sound sensor for recording respiration during sleep (Experimental): PneaVoX sensor, CIDELEC
  Interventions: Device: Sleep apnea diagnosis

INTERVENTIONS:
Device: Sleep apnea diagnosis — Split-night

SUMMARY:
Split-night prospective monocentric study to evaluate, in real conditions, the effectiveness of a disposable tracheal sound sensor.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected obstructive sleep apnea

Exclusion Criteria:

* Lung infection
* Insomnia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2022-04-28 (Estimated); Study Completion 2022-04-28 (Estimated)

PRIMARY OUTCOMES:
Analyzable signal time | One night
  Percentage of the analyzable signal duration compared to the total recorded signal duration